CLINICAL TRIAL: NCT05161897
Title: Individualized Nutrition Therapy for Preventing or Delaying Onset of Type-2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Raedeh Basiri, Assistant Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1825534-1
Record Dates: First submitted 2021-11-02; First posted 2021-12-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes; Cardiovascular Diseases
MeSH Terms: conditions — Prediabetic State; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This arm will receive generalized nutrition therapy throughout the study.
  Participants will receive dietary recommendations based on their needs and will be educated about the recommended amount of carbohydrates for each meal and the carbohydrate choices. Participants will also be provided with a CGM device; however, participants will be blind to the CGM recordings until the end of the study.
- Intervention Group (Experimental): This arm will receive both individualized nutrition therapy and generalized nutrition therapy throughout the study.
  Participants will receive dietary recommendations based on their needs and will be educated about the recommended amount of carbohydrates for each meal and the carb choices. Participants will also be provided with a CGM device and will be educated to review their blood glucose measurements and record above range measures along with time, types and amount of food items consumed, cooking method, and any type of physical activity within one hour before or after the meal. This information will be reviewed by one of the research staff at each visit and will be used to set individualized goals for modifying diet and controlling blood glucose. Participants will visit every 10 days for 30 days to conduct measurements, replace their CGM, set new goals based on their food diary and CGM recordings, and receive further dietary recommendations.
  Interventions: Other: Individualized Nutrition Therapy

INTERVENTIONS:
Other: Individualized Nutrition Therapy — Explained in arm/group description.
  Arms: Intervention Group

SUMMARY:
The overall aim of this feasibility study is to conduct a randomized, controlled intervention providing adults with prediabetes either an individualized nutrition therapy (INT) intervention that contains individualized dietary goal-setting components, the goal being to improve blood glucose, reduce CVD risk factors, and therefore postpone the onset of diabetes and related cardiovascular disease, or standard-of-care generalized dietary recommendation (SOC). The hypothesis is that the INT arm will experience greater benefits in some or all of the following primary outcome variables: improvement in postprandial blood glucose, oral glucose tolerance test, fasting insulin, and calculated insulin sensitivity (HOMA) in individuals with prediabetes. Secondary outcome variables are improved markers of inflammation, antioxidant status, blood lipids, blood pressure, and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45-65 years
* Any race or ethnicity
* Those who have or may have pre-diabetes (will be screened to confirm)
* HbA1c level between 5.7%-6.4% (will be screened to confirm)
* BMI between 25 and 39.9 kg/m2
* Taking stable doses of antihypertensive and/or cholesterol-lowering medications for 3 months or more prior to being enrolled in the study

Exclusion Criteria:

* Pregnant or lactating
* Individuals outside of the HbA1c and BMI inclusion ranges
* Those with active cancer, thyroid, kidney, liver, and pancreatic diseases
* Heavy cigarette smokers (25 cigarettes per day or more)
* Heavy drinkers (>12 alcoholic drinks per week on average)
* Taking more than one hypoglycemic agent (blood sugar lowering medications)
* Having major dietary restrictions
* Participating in any weight loss or dietary program/taking prescribed appetite suppressants
* Participating in another investigational study at the same time as this study
* Anyone who refuses to follow dietary recommendations
* Anyone who refuses to wear the continuous glucose monitoring device as instructed
* Anyone who will not fill out their food dairy and automated self-administered dietary assessment tool

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Change in interstitial glucose concentrations [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Evaluating change in 24hr interstitial glucose concentrations and glycemic variability from baseline measure using a Continuous Glucose Monitoring (CGM) device
Change in insulin sensitivity [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in insulin sensitivity from baseline measure will be assessed using the homeostatic model of insulin resistance (HOMA-IR) and insulin secretion (HOMA-β)
Change in glucose tolerance [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in glucose tolerance from baseline measures will be assessed using an oral glucose tolerance test

SECONDARY OUTCOMES:
Change in inflammation status [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  As assessed by change in blood concentration of c-reactive protein (CRP)
Change in lipid profiles [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  As assessed by change in blood concentration of total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and oxidized LDL (ox-LDL)
Change in markers of endothelial function [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  As assessed by blood concentrations of nitric oxide (NO) and endothelin-1 (ET-1)
Change in blood pressure [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in blood pressure from baseline measures as assessed by measuring resting blood pressure
Change in atherogenic risk ratios [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in atherogenic risk ratios from baseline measures as assessed by (AIP) = Log (TG/HDL-C), CRI-I(TC/HDL-C), CRI-II(LDL-C/HDL-C), AC(TC-HDL-C/HDL-C)
Change in antioxidant status [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in antioxidant status from baseline measure as assessed by measuring total antioxidant capacity (TAC) in blood
Change in dietary intake [Time Frame: baseline, 10 days, 20 days, and 30 days] | baseline, 10 days, 20 days, and 30 days
  Change in dietary intake from baseline measures using data from ASA24 survey for one day in each time frame

CONTACTS AND LOCATIONS:
Overall Officials: Raedeh Basiri, PhD, Principal Investigator — George Mason University
Locations (1):
- Population Health Center Clinic George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No